CLINICAL TRIAL: NCT00140907
Title: A Double-Blind, Randomized, Placebo Controlled Study to Evaluate the Renal Protective Effects of Losartan in Patients With Renal Transplant
Brief Title: ALLOGRAFT, A Study to Evaluate the Renal Protective Effects of Losartan (0954-222)(COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0954-222; MK0954-222; 2005_053
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: High Blood Pressure
MeSH Terms: conditions — Hypertension | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: Placebo
- 2 (Active Comparator): Losartan
  Interventions: Drug: losartan potassium

INTERVENTIONS:
Drug: losartan potassium — 25 mg of oral losartan once daily, with an up-titration to 50 mg of losartan once daily in later visits if serum creatinine did not increase more than 25%. Patients take medication in the morning.
  Arms: 2
Drug: Comparator: Placebo — 25 mg of oral placebo once daily, with an up-titration to 50 mg placebo once daily in later visits if serum creatinine did not increase more than 25%. Patients take medication in the morning.
  Arms: 1

SUMMARY:
To demonstrate that losartan (+ conventional therapy) compared to placebo (+ conventional therapy) will reduce the number of RT patients who experience histological lesions of chronic allograft nephropathy

ELIGIBILITY:
Inclusion Criteria:

* Patients With End Stage Chronic Renal Failure, Four To Eight Week After Receiving A First Or A Second Renal Transplant From A Dead Donor. In The Case Of A Second Transplant The Survival Of The First Graft Must Has Been 6 Month Or More
* Patients Must Have A Serum Creatinine * 2 At Visit 1 And 2. Results Must Be Within 25% Of Each Other. The Baseline Period May Be Extended Until Four More Weeks To Obtain An Additional Serum Creatinine If One Of The First Two Serum Creatinine Results Do Not Qualify
* Patients With Hypertension Must Have A Sitting Blood Pressure < 200/110 Mmhg At The Time Of Randomization
* Normotensive Patients Must Have A Sitting Systolic Blood Pressure >100 Mmhg At The Time Of Randomization

Exclusion Criteria:

* Hyperimmunized Patients At The Transplant Time Or In The Previous 6 Month, With A Pra of 50 %
* Patients With Evidence Of Advanced Liver Disease
* Serum Potassium <3.5 Or >5.5 Meq/L
* History Of Allergy To Losartan
* Other Factors Which May Affect Participation (E.G., Significant Concurrent Or Life Limiting Disease Such As Cancer In The Last Five Year Except Skin Neoplasias, Mental Or Legal Incapacitation, Drug Or Alcohol Abuse Within The Last 2 Years, Extensive Travel Planned In The Next 3 Years, Investigative Drug Trial Within The Last 4 Weeks)
* Patients With Disseminated Or Localized Active Infectious Disease, At The Time Of Transplant
* Acute Graft Rejection In The Grade III Of Banff Classification
* Patients With Double-Transplant (Reno-Pancreatic)
* Patients With Heart Failure Or History Of Myocardial Infarction Requiring Ace Inhibitor Or Aiia Therapies. Presence Or Known History Of Hemodynamically Significant Obstructive Valvular Disease Or Hypertrophic Cardiomyopathy
* Renal Graft Artery Stenosis. An Eco-Doppler Test Must Be Performed In Order To Exclude A Graft Artery Stenosis
* Pregnant Or Nursing Women
* Chronic Use Of Nsaids
* Major Psychotropic Agents Such As Phenothiazines Are Not Permitted, Use Of Lithium Is Not Permitted

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2000-03-14 (Actual); Primary Completion 2005-01-01 (Actual); Study Completion 2005-01-01 (Actual)

PRIMARY OUTCOMES:
Incidence of chronic allograft nephropathy | 24 months post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Natale P, Mooi PK, Palmer SC, Cross NB, Cooper TE, Webster AC, Masson P, Craig JC, Strippoli GF. Antihypertensive treatment for kidney transplant recipients. Cochrane Database Syst Rev. 2024 Jul 31;7(7):CD003598. doi: 10.1002/14651858.CD003598.pub3. PMID 39082471